CLINICAL TRIAL: NCT05546242
Title: A Phase 3b Randomised, Multicentre, Open-label Study Evaluating the Effectiveness of Switching to Two-monthly Long-acting Injectable Cabotegravir and Rilpivirine from First-line Oral Antiretroviral Therapy in HIV-1 Positive Virologically Suppressed Adults with a History Of, or At Risk Of, Sub-optimal HIV Control in Sub-Saharan Africa
Brief Title: Improving HIV-1 Control in Africa with Long Acting Antiretrovirals
Acronym: IMPALA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MRC/UVRI and LSHTM Uganda Research Unit (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMC278LAHTX3005
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — cabotegravir; Rilpivirine; Anti-Retroviral Agents; dolutegravir

STUDY DESIGN:
Intervention Model Description: parallel open-label phase 3b study. Participants will be randomised to continuing current therapy or switching to injectable therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CAB LA + RPV LA Arm (Experimental): The first 4 weeks of the treatment differ depending on whether participant opts for direct to injection (DTI) or Oral lead-in (OLI).
  DTI: participants will remain on daily oral ART for 4weeks after randomization and will receive the 1st injection of IM CAB LA 600mg+RPV LA 900mg at the Month 1 visit. 2nd injections administered at Month 2, followed by maintenance injections every 2 months (Q2M)
  OLI: participants will receive the study intervention in 2 phases:
  1. Participants will receive CAB 30mg+RPV 25mg OD for 4weeks to be taken daily with food. The purpose of the optional OLI Phase is to allow an opportunity for participants to assess tolerability of the combination prior to administration of the injectables. There is no proven benefit to this approach
  2. After 4weeks participants return for the Month 1 visit to receive the 1st IM CAB LA 600mg+RPV LA 900mg injections. The 2nd injections administered at Month 2 and then continuation injections will be administered Q2M
  Interventions: Drug: Cabotegravir/Rilpivirine
- ART Group (Active Comparator): Participants will take a daily oral combination of 2 NRTIs plus DTG 50mg. Ideally, the single tablet fixed-dose combination regimen of (tenofovir disoproxil fumarate [TDF] 300 mg + lamivudine [3TC] 300 mg (or emtricitabine [FTC] 200 mg) + DTG 50 mg) will be used as per local country guidelines up to Month 24. If there are preexisting reasons why TDF or 3TC cannot be used as the NRTI backbone then alternative NRTIs are acceptable. Participants will be permitted to switch daily oral ART drugs in case of toxicity, after discussion with the coordinating center.
  Interventions: Drug: Antiretroviral

INTERVENTIONS:
Drug: Cabotegravir/Rilpivirine — injectable long-acting cabotegravir 600mg + long-acting rilpivirine 900mg administered every 2 months
  Other Names: Vocabria/Rekambys
  Arms: CAB LA + RPV LA Arm
Drug: Antiretroviral — Oral antiretroviral therapy in the form of 2NRTIs + dolutegravir 50mg administered daily
  Other Names: 2NRTIs + dolutegravir 50mg once daily
  Arms: ART Group

SUMMARY:
IMPALA is a randomized, open-label, multicenter, interventional study of 540 virologically suppressed HIV-1 infected adults who have a history of sub-optimal adherence to daily oral ART and/or engagement in HIV care. The study will seek to demonstrate non-inferior antiviral effectiveness of the 2-monthly long-acting injectable combination of cabotegravir/rilpivirine as compared to continuation of first line oral antiretroviral therapy.

DETAILED DESCRIPTION:
IMPALA is a randomized, open-label, multicenter, interventional study of 540 virologically suppressed (<200 c/mL) HIV-1 infected adults (18 years or older) who have a history of sub-optimal adherence to daily oral ART and/or engagement in HIV care. IMPALA seeks to demonstrate the non-inferior antiviral effectiveness of switching to long acting injectable rilpivirine (RPV LA) plus long acting injectable cabotegravir (CAB LA) given every 2 months (Q2M CAB LA + RPV LA) by IM compared to the continuation of first-line daily oral ART containing 2 nucleoside reverse transcriptase inhibitor (NRTIs) plus an integrase strand transfer inhibitor (INSTI; dolutegravir [DTG]).

After providing written informed consent, participants will be evaluated for eligibility during the screening period. Participants who are viremic (HIV VL >200 c/mL) at the time of screening will be virologically suppressed (for >3 months) on a regimen of 2 NRTIs plus DTG prior to randomization. On Day 1 virologically suppressed (<200 c/mL for at least 3 months) individuals will be randomized 1:1 to either continue daily oral ART (2 NRTI + DTG, control arm), or switch to Q2M CAB LA + RPV LA IM, the intervention arm. Those randomized to the intervention arm will be offered either optional oral lead-in (OLI) of 1 month daily oral CAB and RPV or a direct to injection (DTI) approach. This decision to dose with or without an OLI Phase will be determined by the study participant following the informed consent discussion with the investigator. The total duration of the study will be 24 months. Any participant who has received at least a single dose of CAB LA + RPV LA and discontinues the regimen for any reason before Month 24 must start suppressive daily oral ART within 2 months of the last injection. There will be an optional real-world extension phase, provided the regimen is deemed to be non-inferior at Month 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and above
2. HIV-1 infection confirmed in clinic records or by study team.
3. Two consecutive HIV-1 VL <200 copies/mL ≥3 months apart prior to randomization.
4. On an oral regimen of 2NRTI + DTG as part of first line ART
5. Is identified as a participant with a history of, sub-optimal ART adherence or engagement in care based on one or more of the following criteria:

   1. Documented detectable HIV-1 VL (>1000 c/mL) on all-oral ART (EFV/NVP or DTG-based) in the prior 2 years despite being ART-experienced for

      ≥3 months.
   2. History of being lost to follow-up from care (>4 weeks elapsed since a missed scheduled clinic appointment or refill in the prior 2 years).
   3. Failed to link to HIV care despite ≥3 months elapsed since HIV diagnosis.
6. Females: human chorionic gonadotrophin (HCG) negative and willing to use one highly effective form of contraception if woman of reproductive potential
7. Must sign informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study.
8. Willing and able to attend all clinic appointments.

Exclusion Criteria:

1. Not virologically suppressed (VL<200 c/mL) for ≥3 months at the end of the screening process.
2. Previous use, or intention to use, protease inhibitor-based ART at any time.
3. Evidence of prior HIV-1 resistance test with NNRTI drug resistance mutations (other than K103N) and/or INSTI drug resistance mutations.
4. Unwillingness to receive 2 injections on a 2 monthly basis.
5. Unwilling to use a form of contraception.
6. Pregnant, breastfeeding or planning to become pregnant during the study period.
7. Requires tuberculosis therapy or other drug with clinically relevant drug interaction
8. High risk of seizures, including participants with an unstable or poorly controlled seizure disorder.
9. Has active TB or other mycobacterial disease and requires treatment.
10. Advanced liver disease, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or history of cirrhosis.
11. Chronic Hepatitis C with planned or anticipated use of Hep C therapy
12. Evidence of hepatitis B virus (HBV) infection based on the results of testing at Screening for Hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HBcAb), Hepatitis B surface antibody (HBsAb) as follows:

    * Participants positive for HBsAg are excluded
    * Participants negative for HBsAg but positive for HBcAb, with no evidence of HBsAb are excluded NOTE: Participants positive for HBcAb due to prior infection (negative HBsAg status) and with evidence of HBsAb have some immunity to HBV and have low risk of reactivation so are not excluded.
13. Current or anticipated need for chronic anticoagulation therapy.
14. Previous use of oral or injectable CAB or RPV.
15. Any Grade 4 laboratory abnormality at the conclusion of screening process.
16. Creatinine clearance (CrCl) <50 mL/min/1.732 by Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation.
17. Alanine aminotransferase (ALT) > 3×upper limit of normal (ULN).
18. Has a tattoo or other dermatological condition overlying the gluteus region that may interfere with interpretation of ISRs.
19. Has ongoing or clinically significant medical conditions that in the opinion of the investigator may interfere with the absorption, distribution, metabolism or excretion of the study interventions or could affect participant safety.
20. Has pre-existing physical or mental condition which, in the opinion of the investigator, may interfere with the participant's ability to comply with the dosing schedule and/or protocol evaluations or which may compromise the safety of the participant.
21. Known allergies, hypersensitivity, or intolerance to cabotegravir or rilpivirine or its excipients.
22. Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days before the planned first dose of study intervention or is currently enrolled in another interventional study.
23. Has received any prohibited medication listed in Section 6.8.2, Prohibited Medications and Non-drug Therapies and is unwilling or unable to switch to an alternate medication.
24. Has been treated with any of the following agents within 28 days of Screening:

    1. Radiation therapy.
    2. Cytotoxic chemotherapeutic agents.
    3. Tuberculosis therapy with the exception of isoniazid (isonicotinyl hydrazid, INH).
    4. Anticoagulation agents (e.g., warfarin and direct oral anticoagulants).
25. Is using immunomodulators that alter immune responses (such as chronic systemic corticosteroids, interleukins, or interferons). Note: Participants using short-term steroid tapers, topical, inhaled and intranasal corticosteroids, topical imiquimod are eligible for enrolment.
26. Treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening.
27. QTc interval >450 ms (if QTc interval is >450 ms on the ECG read out, then it should be corrected according to Fridericia; https://www.mdcalc.com/corrected-qt-interval-qtc) within 90 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2022-12-08 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
HIV-1 viral load at 12 months | 12 months
  Proportion with plasma HIV-1 viral load (VL) <50 c/mL at 12 months (by Food and Drug Administration [FDA] snapshot algorithm)

SECONDARY OUTCOMES:
Confirmed virologic failure on 2 consecutive occasions | 12 months
  Proportion with confirmed virologic failure (CVF) [plasma HIV-1 VL ≥200 c/mL on 2 consecutive occasions]
Confirmed virologic failure on 2 consecutive occasions | 24 months
  Proportion with confirmed virologic failure (CVF) [plasma HIV-1 VL ≥200 c/mL on 2 consecutive occasions]
Lost to follow up | 12 months
  Proportion with LTFU [>4 weeks elapsed since their last missed appointment]
Lost to follow up | 24 months
  Proportion with LTFU [>4 weeks elapsed since their last missed appointment]
HIV-1 viral load <200c/mL | 12 months
  Proportion with plasma HIV-1 VL <200 c/mL
Virologic response | 12 months and 24 months
  Proportion with plasma HIV-1 VL <50 c/mL
Virologic non-response | 24 months
  Proportion with plasma HIV-1 VL >=50 c/mL (by FDA snapshot algorithm)
Change in CD4+ T cell count | 12 months
  Change in CD4+ T cell count from baseline
Change in CD4+ T cell count | 24 months
  Change in CD4+ T cell count from baseline
HIV disease progression | 24 months
  Incidence of HIV disease progression (HIV/AIDS related hospitalizations, illness or deaths)
Adverse Events | 12 months
  Incidence of adverse events (AEs)
Adverse Events | 24 months
  Incidence of adverse events (AEs)
Grade 3 and 4 Adverse Events | 12 months
  Incidence of AEs, Grade 3 and 4 excluding injection site reactions
Grade 3 and 4 Adverse Events | 24 months
  Incidence of AEs, Grade 3 and 4 excluding injection site reactions
Injection Site Reactions | 24 months
  Frequency of injection site reactions of any grade
Resistance Emergence | 12 months and 24 months
  Frequency of emergence of new integrase strand transfer inhibitor and non-nucleoside reverse transcriptase inhibitor resistance mutations in those who develop virologic failure

OTHER OUTCOMES:
Change in health-related quality of life | 12 months and 24 months
  Change from baseline in EQ-5D-5L
Change in health-related quality of life | 12 months and 24 months
  Change from baseline in MOS-HIV
Change in health-related quality of life | 6 months, 12 months and 18 months
  quality of life outcomes in in-depth interviews
Treatment satisfaction | 12 months and 24 months
  For participants in the CAB LA + RPV LA group, change from baseline in HIVTSQ scores
Treatment preference | 12 months and 24 months
  For participants randomized to the CAB LA + RPV LA group, preference for CAB LA + RPV LA compared to daily oral ART regimen using a single dichotomous preference question
Medical resource utilisation | 24 months
  medical resource utilisation
Medical resource utilisation | 24 months
  Clinic / hospital attendances
Medical resource utilisation | 24 months
  Rates of opportunistic infections and other illnesses
Programmatic acceptability of Q2M CAB LA + RPV LA | 24 months
  Thematic analysis of data from interviews and focus group discussions with participants, healthcare workers and key stakeholders
Treatment adherence | 24 months
  Self-reported adherence and pill count for daily oral ART and delayed/missed injections for CAB LA + RPV LA

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Cresswell, MBChB, PhD, Principal Investigator — MRC/UVRI & LSHTM
Locations (7):
- Kenya (2):
  - Jaramogi Oginga Odinga Teaching & Referral Hospital, Kisumu
  - Kenyatta National Hospital, Nairobi
- South Africa (2):
  - Desmond Tutu Health Foundation, Cape Town
  - CAPRISA, Durban
- Uganda (3):
  - Entebbe Grade A Hospital, Entebbe
  - JCRC Fort Portal, Fort Portal
  - Infectious Diseases Institute, Kampala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tumusiime VB, Ruzagira E, Norcross C, Eshun-Wilsonova I, Kitonsa J, Bahemuka UM, Grint D, Kimbugwe G, Kakande A, Lawrence DS, Mwendia F, Van Solingen R, Van Eygen V, Addo Boateng F, Cresswell F; IMPALA study team. Efficacy and Safety of Long-acting Injectable Cabotegravir and Rilpivirine in Improving HIV-1 Control in sub-Saharan Africa: Protocol for a Phase 3b Open-Label Randomized Controlled Trial (IMPALA). Wellcome Open Res. 2025 Mar 28;10:166. doi: 10.12688/wellcomeopenres.23363.1. eCollection 2025. PMID 41040645